CLINICAL TRIAL: NCT03437915
Title: BrUOG 351: Pre-Operative Accelerated Partial Breast Irradiation (APBI) Using Non-Invasive Image-Guided Breast Brachytherapy (NIBB)
Brief Title: BrUOG 351: PRE-OPERATIVE APBI USING NIBB
Acronym: 351
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Secondary to medicare coverage determination
Sponsor: Jaroslaw Hepel (Other)
Collaborators: Brown University (Other); Rhode Island Hospital (Other); Women and Infants Hospital of Rhode Island (Other)
Responsible Party: Sponsor-Investigator, Jaroslaw Hepel, Principal Investigator: Sponsor-Investigator, Brown University
Organization: Brown University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BrUOG 351
Record Dates: First submitted 2018-02-09; First posted 2018-02-19 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Breast Cancer; Invasive Breast Cancer; Ductal Carcinoma in Situ
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Intraductal, Noninfiltrating | interventions — Mastectomy, Segmental

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment Arm (Experimental): 28.5 Gy delivered in 5 daily fractions then 4-12 weeks post NIBB, surgery via partial mastectomy
  Interventions: Radiation: NIBB: accuboost; Procedure: Partial mastectomy

INTERVENTIONS:
Radiation: NIBB: accuboost — 28.5 Gy delivered in 5 daily fractions
Procedure: Partial mastectomy — 4-12 weeks post NIBB

SUMMARY:
Partial breast irradiation is typically performed after surgical removal of the tumor. Partial breast irradiation allows for focused radiation to the area from which the cancer was removed, sparing breast tissue from the potential bad effects of radiation compared to radiating the whole breast, which was the standard of care for many years. This study is evaluating the use of partial breast irradiation with NIBB performed before surgery instead of after surgery.This should allow researchers to target the cancer even more accurately and result in less normal breast tissue receiving radiation which may cause less side effects and/or a better cosmetic outcome.

In this study partial breast treatment will be given with NIBB in 5 treatments over about 1 week. Surgical removal of the tumor will then be performed between 4-12 weeks following radiation treatment. Researchers believe that participant's risk of complications from surgery will not be higher after getting these radiation treatments than it would have been if participants had surgery first, but that is one of the things researchers are studying.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed histological diagnosis of invasive breast carcinoma and/or DCIS (Invasive lobular carcinoma excluded);
* Age greater or equal to 60 years old;
* Life expectancy > 6 months;
* Candidate for breast conserving surgery who intends to undergo breast conserving surgery as confirmed in writing by treating physician in consultation with surgeon
* Clinically lymph node negative (cN0) as confirmed in writing by patient's treating physician. If patient has suspicious lymphadenopathy on imaging it is required that patient undergo a biopsy to confirm cN0.
* Tumor size by imaging ≤ 2cm; (Tis or T1)
* Estrogen receptor positive if invasive disease (DCIS can be ER negative);
* Her2neu negative if invasive disease;
* Nuclear Grade 1 or 2 if invasive disease (DCIS can be Grade 3);
* ECOG performance status of 0-2 (Appendix 1);
* Informed consent signed.

Exclusion Criteria:

* Excisional biopsy or ipsilateral breast surgery within 6 months;
* Invasive lobular histology;
* Definitive LVSI on biopsy;
* Suspicious imaging findings suggesting multi-focal or multi-centric disease, unless biopsy proven benign;
* Paget's disease of the nipple
* Distant metastases;
* Known BRCA 1/2 Mutation
* Active lupus or scleroderma,;
* Psychiatric or addictive disorder that would preclude attending follow-up;
* Neoadjuvant chemotherapy or endocrine therapy (adjuvant therapy is permitted);
* Breast Implants;
* Tumor not well visualized on AccuBoost imaging;
* Breast separation with compression > 8cm at time of simulation.

Min Age: 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — This study is specifically enrolling female patients with breast cancer age 60 or older.
Enrollment: 0 (Actual)
Dates: Start 2019-03 (Estimated); Primary Completion 2020-01-21 (Actual); Study Completion 2020-01-21 (Actual)

PRIMARY OUTCOMES:
Feasibility of APBI including rate of surgical complications. | Surgery will occur 4-12 weeks post NIBB treatment
Toxicity of pre-op APBI including rate of surgical complications. | Defined at up to 6 weeks post APBI
  Defined as acute (during treatment and through 4 weeks post treatment)
Toxicity of surgical complications | Surgery to occur 4-12 weeks post radiation and post-op complications collected through 3 months post surgery

SECONDARY OUTCOMES:
Assess and report late toxicity | 6 weeks post treatment through 3 years
  Late toxicity defined as 6 weeks post NIBB through 3 years in follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Jaroslaw Hepel, MD, Principal Investigator — Rhode Island Hospital/ BrUOG